CLINICAL TRIAL: NCT04595968
Title: A Randomized, Double Blind Sham Controlled Clinical Trial to Evaluate the Efficacy of Vestibular Nerve Stimulation (VeNS), Together with a Lifestyle Modification Program, Compared to a Sham Control with a Lifestyle Modification Program, As a Means of Improving Glycemic Control in Adults with Type 2 Diabetes Mellitus
Brief Title: Electrical Vestibular Nerve Stimulation (VeNS) Compared to Sham Control As a Means of Improving Glycemic Control in Adults with Type 2 Diabetes Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Neurovalens Ltd. (Industry)
Collaborators: University College Dublin (Other); CS Lifescience (Unknown); Clinical Trial Mentors (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: VeSTALDM01
Record Dates: First submitted 2020-10-12; First posted 2020-10-22 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vestal DM active device (Experimental): 150 subjects randomised to receive active device plus lifestyle intervention for 24 weeks
  Interventions: Device: Vestal DM Active device; Behavioral: Lifestyle modification
- Vestal DM sham device (Sham Comparator): 150 subjects randomised to receive sham device plus lifestyle intervention for 24 weeks.
  Interventions: Behavioral: Lifestyle modification; Device: Vestal DM Sham device

INTERVENTIONS:
Device: Vestal DM Active device — Battery powered non-invasive neurostimulation device
  Arms: Vestal DM active device
Behavioral: Lifestyle modification — Subjects are prescribed a low calorie (500kcal deficit) diet if their BMI is ≥25. If a subject has a BMI of ≤24.9, they will be provided with guidance on ensuring their recommended daily dietary intake is achieved throughout the course of the trial (i.e 2,500kcal/day for men and 2,000kcal/day for women)
Device: Vestal DM Sham device — Placebo comparator sham device (no active stimulation)
  Arms: Vestal DM sham device

SUMMARY:
Trial Title A randomized, double blind sham controlled clinical trial to evaluate the efficacy of vestibular nerve stimulation (VeNS), together with a lifestyle modification program, compared to a sham control with a lifestyle modification program, as a means of improving glycemic control in adults with type 2 diabetes mellitus.

The aim of this study is to evaluate the efficacy of non-invasive electrical vestibular nerve stimulation (VeNS), together with a lifestyle modification program, as a method of reducing HbA1c, as compared to a sham control.

Allocation: Randomized to either active device or control device usage. All subjects will receive the same lifestyle advice.

Endpoint classification: Efficacy Study Intervention Model: Parallel Assignment in 1:1 active to control allocation Trial Participants: Those who have been diagnosed with Type 2 diabetes mellitus.

Planned Trial Period: The study will last 24 weeks in total for each subject. The primary analysis will be conducted at the 24 weeks timepoint.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained before any trial-related activities. Trial-related activities are any procedures that are carried out as part of the trial, including activities to determine suitability for the trial.
* Male or female, age ≥ 22 years and ≤ 70 years at the time of signing informed consent. (At the US sites). The non-US sites will recruit subjects aged ≥ 18 and ≤ 70 years.
* Diagnosed with Type 2 DM ≥ 90 days prior to day of enrolment
* HbA1c (glycated hemoglobin) ≥ 6.5 and ≤ 9.5% (48-80 mmol/mol) (both inclusive).
* If taking medication to treat diabetes, a stable dose of no more than 3 anti-diabetic medications for at least 90 days prior to enrolment.
* BMI ≥ 25 at non-US sites
* Must be under care of physician for follow-up of their type 2 DM (this can be a Primary Care Physician (PCP), endocrinologist or other hospitalist).
* Must agree to continue to participate with their routine diabetes care program.
* Access to Wi-Fi.

Exclusion Criteria:

* Diagnosis of Type 1 diabetes mellitus
* Diagnosis of diabetic neuropathy
* Diagnosis of diabetic nephropathy
* Diagnosis of retinopathy
* Skin breakdown, eczema or other dermatological condition (e.g. psoriasis) affecting the skin behind the ears. Any disorder which in the investigator's opinion might jeopardize subject's safety or compliance with the protocol.
* Taking beta-blockers (if previously then can enroll if off ≥ 30 days).
* Taking insulin (if previously on insulin then should be off for ≥ 90 days prior to enrolment).
* Female who is pregnant, breast-feeding or intends to become pregnant or is of child-bearing potential and not using an adequate contraceptive method (adequate contraceptive measure as required by local regulation or practice)
* History of pancreatitis
* History of pancreatic surgery
* Hemochromatosis
* Either of the following within the previous year: myocardial infarction; or acute coronary syndrome.
* History of stroke
* History of epilepsy
* Splenectomy (due to effect on red blood cell turnover)
* History of anemia (if resolved for > 90 days with treatment then can enroll)
* Blood transfusion within 90 days of enrolment (due to effect on HbA1c). (If transfusion occurs once enrolled then subject will be withdrawn).
* A diagnosis of a hemoglobinopathy (e.g. sickle cell disease and thalassemia, although those with sickle cell or thalassemic trait would be allowed to enroll);
* If on dietary supplements or herbal remedies, then if the subject is taking a preparation that might affect glycemic control they will be excluded. Specifically, subject will be excluded if taking biotin (vitamin B7); alpha-lipoic acid; chromium; herbal preparations marketed as being for diabetes.
* History of being diagnosed with renal, heart or liver failure
* History of active migraines with aura
* History of head injury requiring intensive care or neurosurgery.
* Change in diabetic medication within the last 90 days (prior to enrolment).
* Regular use (more than twice a month) of antihistamine medication within the last 6 months. Note: If the participant is taking Fexofenadine, they can be eligible for the trial. If the participant is on another anti-histamine medication they can voluntarily opt to switch to Fexofenadine and enrol in the trial after a washout period of 2 weeks.
* Current use of H2-receptior antagonist medication? (e.g., cimetidine, famotidine)
* History or presence of malignancy within the last year (except basal and squamous cell skin cancer and in-situ carcinomas)
* A diagnosis of myelofibrosis or a myelodysplastic syndrome.
* Previous use of Modius device
* Participation in other clinical trials sponsored by Neurovalens (e.g. Vestal study)
* Presence of permanently implanted battery powered medical device or stimulator (e.g., pacemaker, implanted defibrillator, deep brain stimulator, vagal nerve stimulator etc.)
* Have a member of the same household who is currently participating in this study.
* History of vestibular dysfunction or other inner ear disease (as assessed on the screening questionnaire)
* Failure to pass the ATMAS Flex hearing test
* Failure to demonstrate a willingness for lifestyle modification (i.e diet and exercise) if BMI is ≥25 (as assessed on the screening questionnaire)
* Failure to agree to weekly engagements with the Clinical Trial Mentors during trial participation
* Failure to agree to use of device daily during trial participation (no more than 2 weeks usage drop without reasonable explanation)
* Use of any medication (e.g. hormonal modulators or corticosteroids) that could cause iatrogenic T2DM. (NB Topical steroid use is acceptable if judged by PI to be unrelated).
* Any other medical condition, or medication use, that in the opinion of the PI/CI is likely to make the subject refractory to VeNS.

Ages: 22 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 267 (Actual)
Dates: Start 2021-05-21 (Actual); Primary Completion 2024-08-06 (Actual); Study Completion 2024-08-06 (Actual)

PRIMARY OUTCOMES:
Change in glycated hemoglobin (HbA1c) | 24 weeks
  Change in HbA1c levels over the course of the study
Frequency of all device related Serious Adverse Events | 24 weeks
  Frequency of all Device Related Serious Adverse Events (SAEs).

SECONDARY OUTCOMES:
Participants who achieve HbA1c targets | 24 weeks
  1. Participants Who Achieve HbA1c < 7.0 % (53 mmol/Mol) ADA Target (Yes/no),
  2. Participants Who Achieve ≥ 0.5% HbA1c reduction (Performance goal of ≥ 50% of active group to be specified in SAP)
  3. Participants Who Achieve HbA1c ≤ 6.5 % (48 mmol/Mol) AACE Target (Yes/no)
Change in Body weight | 24 weeks
  Change in body weight as a percentage
Reduction of HbA1c in relation to weight loss | 24 weeks
  Assessment of reduction in HbA1c (%) per kg weight lost.
Change in BMI | 24 weeks
  Change in BMI across the duration of the study
Change in waist-hip ratio (WHR) | 24 weeks
  Change in waist-hip ratio (WHR) over time
Change in body composition (DXA scan) | 24 weeks
  Change in body composition (body fat percentage; body fat mass; visceral fat; muscle mass; bone mass) measured via a DXA scan
Change in atherogenic index | 24 weeks
  Change in the atherogenic index (ratio of total cholesterol to High Density Lipoprotein (HDL)
Change in Total Cholesterol | 24 weeks
  Change in Total Cholesterol over time
Change in High Density Lipoprotein (HDL) | 24 weeks
  Change in High Density Lipoprotein (HDL) over time
Change in Low Density Lipoprotein (LDL) | 24 weeks
  Change in Low Density Lipoprotein (LDL) over time
Change in Triglycerides | 24 weeks
  Change in Triglycerides over time
Change in Very-low-density lipoprotein (VLDL) | 24 weeks
  Change in Very-low-density lipoprotein (VLDL) over time
Change in pulse rate | 24 weeks
  change in pulse rate over time
Change in Mean arterial pressure (MAP) | 24 weeks
  Change in Mean arterial pressure (MAP). (MAP is approximately equal to (2/3 x DBP) + (1/3 x SP))
Change in fasting plasma glucose | 24 weeks
  Change in fasting plasma glucose
Change in 7 point Self Measured Blood Glucose (SMBG) | 24 weeks
  Change in 7 point SMBG - Ratio to Baseline
Change in anti-diabetic medication | 24 weeks
  Change in anti-diabetic medication. Diabetic medications will be summarized in terms of an increase, decrease or no change in medication, by treatment group. This assessment will be made by suitably qualified members of the study team.
Change in cardiovascular medication | 24 weeks
  Change in cardiovascular medication. The changes in cardiovascular medications will be summarized in terms of an increase, decrease or no change in cardiovascular medication, by treatment group. This assessment will be made by suitably qualified members of the study team.
Change in audit of diabetes dependent Quality of Life (QoL) score | 24 weeks
  Change in Audit of Diabetes Dependent Quality of Life Total Score (ADDQoL)
Tolerability of treatment | 24 weeks
  Tolerability of treatment summarized by:
  Duration of Exposure Device usage data Mentor support group usage (hours per week)
Change in healthcare resource use | 24 weeks
  Change in healthcare resource use over time
Change in Diabetes Treatment Satisfaction Questionnaire (DTSQ) | 24 weeks
  Change in Diabetes Treatment Satisfaction Questionnaire (DTSQ) score over time
Change in EQ-5D-5L | 24 weeks
  Change in EQ-5D-5L quality of life score over time
Frequency of Adverse Events (AEs) | 24 weeks
  Frequency of Adverse Events (AEs) (including Serious Adverse Events (SAEs)).
Frequency of hypoglycemic episodes | 24 Weeks
  Change from baseline
Frequency of episodes resulting with HbA1c > 10% | 24 weeks
  Change from baseline
Change in hearing by means of AMTAS flex device | 24 weeks
  Change from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Erik Viirre, MD PhD, Principal Investigator — UC San Diego
Locations (16):
- United States (15):
  - University of Alabama, Birmingham, Alabama
  - UC San Diego, Exercise and Physical Activity Resource Center, La Jolla, California
  - Northern California Research, Sacramento, California
  - New Med Research, Hollywood, Florida
  - South Florida Research Organization, Medley, Florida
  - Adult Medicine of Lake County, Mt. Dora, Florida
  - Oviedo Medical Research, Oviedo, Florida
  - ActivMed Practices & Research, Methuen, Massachusetts
  - Billings Clinic, Billings, Montana
  - Palm Research Center, Las Vegas, Nevada
  - ActivMed Practices & Research, Portsmouth, New Hampshire
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Complete Health Partners, Nashville, Tennessee
  - Biopharma Informatic, McAllen, Texas
  - Charlottesville Medical Research Center, Charlottesville, Virginia
- St. Vincent's University Hospital, Dublin, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: Undecided